CLINICAL TRIAL: NCT00571844
Title: Behavioral Treatment of High Blood Pressure
Brief Title: ENCORE: Exercise and Nutritional Interventions for Cardiovascular Health
Acronym: ENCORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00007858; 5R01HL074103 (NIH); 4842 (Other: Duke legacy protocol number)
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Exercise; Diet; Biomarkers
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DASH diet (Experimental)
  Interventions: Behavioral: DASH diet
- DASH diet plus Weight loss (Experimental)
  Interventions: Behavioral: DASH diet plus Weight loss
- Usual Care (No Intervention): Usual Care Control Group: Patients in the Usual Care control group will be asked to maintain their usual dietary and exercise habits for 4 months until they are re-evaluated. At biweekly intervals we will ask patients to describe any spontaneous changes in their eating habits or food preferences. To ensure patient safety, BPs will also be monitored biweekly by our staff.

INTERVENTIONS:
Behavioral: DASH diet — Participants in the DASH diet condition receive instruction in modifying the content of their diet to meet DASH guidelines. Participants are explicitly asked not to exercise or to attempt weight loss at this time, and to focus their attention on what they eat. Following the 2-week feeding period, participants will receive instruction on the DASH diet and feedback on their adherence to the diet in a series of half-hour, weekly small group sessions (3 to 5 participants).
  Arms: DASH diet
Behavioral: DASH diet plus Weight loss — Participants in the DASH diet plus weight loss condition will receive the DASH dietary intervention as described in the DASH diet intervention and will participate in a program to promote weight loss consisting of 2 components: Supervised Aerobic Exercise and CBWL (Cognitive Behavioral Weight loss). During supervised exercise participants will exercise 3x/week under medical supervision at the Duke Center for Living. A trained exercise physiologist will supervise all exercise sessions, and will obtain exercise BP measurements to make sure that BP is not abnormally elevated. For the CBWL participants will meet in small groups of 3-5 patients for instruction in weight management techniques. CBWL will include Appetite Awareness Training (AAT), a self-monitoring strategy developed to provide more specific guidelines regarding how much to eat. Individuals learn to identify moderate hunger and fullness and use these internal cues to guide their eating.
  Arms: DASH diet plus Weight loss

SUMMARY:
This study is an NIH-funded clinical trial conducted at Duke Medical Center evaluating the effects of the DASH diet alone and combined with a behavioral weight loss program on blood pressure and various vascular measures. Eligible patients must be unmedicated with blood pressure values ranging from approximately 130/85 to 159/99. Our primary hypothesis are as follows: (1) The DASH diet alone and combined with a behavioral weight management program will result in greater BP reductions than Usual Care controls at the end of the 4 month treatment period; (2) The DASH diet in combination with a behavioral weight management program will be more effective in lowering BP than the DASH diet alone; (3) The DASH diet alone and the DASH diet combined with the behavioral weight management program will result in greater improvements in cardiac, metabolic, and vascular function compared to the control condition; and (4) The combined DASH diet and weight management intervention also will be the most effective treatment in maintaining BP reductions at 1-year follow-up.

DETAILED DESCRIPTION:
The present application seeks to extend previous findings by a) evaluating the efficacy of the DASH diet in a free-living situation; (b) considering the DASH diet alone and in combination with a behavioral weight loss program including aerobic exercise; (c) examining the impact of diet and exercise on cardiac, metabolic, and vascular function, including measures of arterial stiffness, endothelial function, baroreflex control, body composition, insulin resistance, cardiac hemodynamics, and left ventricular (LV) geometry and mass; and (d) following patients for one year to determine the longer term impact of the interventions on BP, body weight, and cardiovascular function.

ELIGIBILITY:
Inclusion Criteria:

1. Baseline SBP 130-159 mmHg (+/- 2mmHg) or DBP 85-99 mmHg (+/- 2 mm Hg)
2. Age 35 years or older
3. BMI 25.0-39.99 kg/m², with a maximum weight of 300 lbs
4. Willing and able to participate fully in all aspects of the intervention
5. Must currently be sedentary (less than 3x/wk for 30 mins each time)
6. Informed consent

Exclusion Criteria:

1. Use of weight-loss medication and/or participation in a structured weight- loss program in the 3 months prior to 1st screening visit.
2. Regular use of an anti-hypertensive drug or other drugs that raise or lower BP and if discontinued use, must be off for 1 month before screening
3. Current use of insulin or oral hypoglycemic agents
4. Current use of medications for treatment of psychosis or manic-depressive illness.
5. ADHD medications (Ritalin/Aderol/amphetamines
6. Cardiovascular Event
7. Coronary Artery Disease
8. Congestive Heart Failure
9. Current symptoms of Angina for peripheral vascular disease
10. Cancer diagnosis (except for non-melanoma skin cancer) or treatment in past 2 years
11. Fasting blood sugar >126 mg/dl
12. Gastric Bypass/Bariatric Surgery
13. Pyschiatric hospitalization in the past 2 years.
14. Unable or willing to consume all of the dietary foods provided during the 2-week feeding.
15. Consumption of more than 21 alcoholic drinks per week or binge drinking
16. Alcoholism as determined by the Alcohol AUDIT (screening questionnaires)
17. Planning to leave the area prior to the anticipated end of participation
18. Body weight change of >15lbs in the 3 months prior to the 1st screening visit
19. Pregnant, breast feeding, or planning pregnancy prior to end of participation
20. Current participation in another clinical trial until after completion of T2
21. Investigator discretion for safety or adherence reasons
22. Controlled substance abuse

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2003-10; Primary Completion 2009-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 4 months

SECONDARY OUTCOMES:
Ambulatory blood pressure,vascular function,left ventricular geometry, glucose tolerance,body composition, quality of life | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: James A. Blumenthal, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Background] Svetkey LP, Harsha DW, Vollmer WM, Stevens VJ, Obarzanek E, Elmer PJ, Lin PH, Champagne C, Simons-Morton DG, Aickin M, Proschan MA, Appel LJ. Premier: a clinical trial of comprehensive lifestyle modification for blood pressure control: rationale, design and baseline characteristics. Ann Epidemiol. 2003 Jul;13(6):462-71. doi: 10.1016/s1047-2797(03)00006-1. PMID 12875806
- [Background] The sixth report of the Joint National Committee on prevention, detection, evaluation, and treatment of high blood pressure. Arch Intern Med. 1997 Nov 24;157(21):2413-46. doi: 10.1001/archinte.157.21.2413. PMID 9385294
- [Background] Blumenthal JA, Sherwood A, Gullette EC, Babyak M, Waugh R, Georgiades A, Craighead LW, Tweedy D, Feinglos M, Appelbaum M, Hayano J, Hinderliter A. Exercise and weight loss reduce blood pressure in men and women with mild hypertension: effects on cardiovascular, metabolic, and hemodynamic functioning. Arch Intern Med. 2000 Jul 10;160(13):1947-58. doi: 10.1001/archinte.160.13.1947. PMID 10888969
- [Background] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655
- [Background] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Background] Blumenthal JA, Sherwood A, Gullette EC, Georgiades A, Tweedy D. Biobehavioral approaches to the treatment of essential hypertension. J Consult Clin Psychol. 2002 Jun;70(3):569-89. PMID 12090370
- [Background] Linden W, Chambers L. Clinical effectiveness of non-drug treatment for hypertension: a meta-analysis. Ann Behav Med. 16:35-45, 1994.
- [Background] Jeffery RW. Weight management and hypertension. Ann Behav Med. 13:18-22, 1991.
- [Background] Windhauser MM, Evans MA, McCullough ML, Swain JF, Lin PH, Hoben KP, Plaisted CS, Karanja NM, Vollmer WM. Dietary adherence in the Dietary Approaches to Stop Hypertension trial. DASH Collaborative Research Group. J Am Diet Assoc. 1999 Aug;99(8 Suppl):S76-83. doi: 10.1016/s0002-8223(99)00420-4. PMID 10450298
- [Background] Svetkey LP, Simons-Morton D, Vollmer WM, Appel LJ, Conlin PR, Ryan DH, Ard J, Kennedy BM. Effects of dietary patterns on blood pressure: subgroup analysis of the Dietary Approaches to Stop Hypertension (DASH) randomized clinical trial. Arch Intern Med. 1999 Feb 8;159(3):285-93. doi: 10.1001/archinte.159.3.285. PMID 9989541
- [Background] Hinderliter A, Sherwood A, Gullette EC, Babyak M, Waugh R, Georgiades A, Blumenthal JA. Reduction of left ventricular hypertrophy after exercise and weight loss in overweight patients with mild hypertension. Arch Intern Med. 2002 Jun 24;162(12):1333-9. doi: 10.1001/archinte.162.12.1333. PMID 12076231
- [Background] Blumenthal JA, Siegel WC, Appelbaum M. Failure of exercise to reduce blood pressure in patients with mild hypertension. Results of a randomized controlled trial. JAMA. 1991 Oct 16;266(15):2098-104. PMID 1920698
- [Derived] Hinderliter AL, Smith P, Sherwood A, Blumenthal J. Lifestyle Interventions Reduce the Need for Guideline-Directed Antihypertensive Medication. Am J Hypertens. 2021 Oct 27;34(10):1100-1107. doi: 10.1093/ajh/hpab090. PMID 34107031
- [Derived] Hinderliter AL, Sherwood A, Craighead LW, Lin PH, Watkins L, Babyak MA, Blumenthal JA. The long-term effects of lifestyle change on blood pressure: One-year follow-up of the ENCORE study. Am J Hypertens. 2014 May;27(5):734-41. doi: 10.1093/ajh/hpt183. Epub 2013 Oct 1. PMID 24084586
- [Derived] Epstein DE, Sherwood A, Smith PJ, Craighead L, Caccia C, Lin PH, Babyak MA, Johnson JJ, Hinderliter A, Blumenthal JA. Determinants and consequences of adherence to the dietary approaches to stop hypertension diet in African-American and white adults with high blood pressure: results from the ENCORE trial. J Acad Nutr Diet. 2012 Nov;112(11):1763-73. doi: 10.1016/j.jand.2012.07.007. Epub 2012 Sep 19. PMID 23000025
- [Derived] Blumenthal JA, Babyak MA, Sherwood A, Craighead L, Lin PH, Johnson J, Watkins LL, Wang JT, Kuhn C, Feinglos M, Hinderliter A. Effects of the dietary approaches to stop hypertension diet alone and in combination with exercise and caloric restriction on insulin sensitivity and lipids. Hypertension. 2010 May;55(5):1199-205. doi: 10.1161/HYPERTENSIONAHA.109.149153. Epub 2010 Mar 8. PMID 20212264
- [Derived] Blumenthal JA, Babyak MA, Hinderliter A, Watkins LL, Craighead L, Lin PH, Caccia C, Johnson J, Waugh R, Sherwood A. Effects of the DASH diet alone and in combination with exercise and weight loss on blood pressure and cardiovascular biomarkers in men and women with high blood pressure: the ENCORE study. Arch Intern Med. 2010 Jan 25;170(2):126-35. doi: 10.1001/archinternmed.2009.470. PMID 20101007